CLINICAL TRIAL: NCT02590003
Title: A Randomized Phase II Trial of Combination Versus Single Agent Chemotherapy in High-risk Elderly Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Single Agent Versus Combination Chemotherapy to Treat High-risk Elderly With Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial was stopped after non-response to treatment.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1403013529
Record Dates: First submitted 2015-10-12; First posted 2015-10-28 (Estimated); Results first posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-01

CONDITIONS: Carcinoma, Non-small Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platinum-based doublet chemotherapy (Experimental): * Carboplatin AUC 5 30 minute infusion IV on day 1
  * Nab-paclitaxel 100mg/mg2 30 minute infusion IV on days 1, 8 of a 21 day cycle
  Interventions: Drug: Carboplatin; Drug: Nab-paclitaxel
- Single agent chemotherapy (Active Comparator): -Nab-paclitaxel 100mg/mg2 30 minute infusion IV on days 1, 8 of a 21 day cycle
  Interventions: Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Carboplatin
  Arms: Platinum-based doublet chemotherapy
Drug: Nab-paclitaxel

SUMMARY:
This study will enroll elderly patients with advanced non-small cell lung cancer who are at high risk of developing chemotherapy toxicity (side effects). Patients will receive treatment with either a platinum-based doublet chemotherapy with carboplatin/nab-paclitaxel or single agent nab-paclitaxel of chemotherapy. Response to treatment and treatment toxicity will be compared in the two treatment groups to determine the best treatment strategy for this group of patients.

DETAILED DESCRIPTION:
The primary objective of this trial is to compare the treatment failure-free survival rate in high-risk elderly patients, identified by geriatric assessment, treated with either a platinum-based doublet chemotherapy with carboplatin/nab-paclitaxel or single agent nab-paclitaxel in advanced non-small cell lung cancer. Treatment failure-free survival is the most appropriate primary outcome as it captures excessive toxicity due to chemotherapy in addition to death and disease progression.

The secondary objectives are to evaluate grade 3-5 toxicities, overall response rate, progression free survival, symptom assessment, and overall survival between the two randomization arms.

ELIGIBILITY:
Inclusion Criteria:

1. Patient able and willing to comply with study procedures as per protocol, including the geriatric assessment at the time of study enrollment.
2. Patient able to understand and willing to sign and date the written voluntary informed consent form (ICF) at screening visit prior to any protocol-specific procedures.
3. Patients must have histological or cytological confirmed primary non-small cell lung cancer (adenocarcinoma, large cell carcinoma, squamous, or unspecified). Disease must be stage IV Non-Small Cell Lung Cancer (NSCLC). Disease may be either newly diagnosed or recurrent after previous surgery and/or irradiation. Primary or metastatic site for biopsy is allowed
4. Patients may have measurable or non-measurable disease documented by CT or MRI. The CT from a combined PET/CT may be used to document only non-measurable disease. Measurable disease must be assessed within 30 days prior to registration per response evaluation criteria in solid tumors (RECIST) v1.1. Pleural effusions, ascites and laboratory parameters are not acceptable as the only evidence of disease. Non- measurable disease must be assessed within 30 days prior to registration. All disease must be assessed and documented on the Baseline Tumor Assessment Form.
5. Prior chemotherapy for curative intent is permitted providing the cytotoxic chemotherapy was completed ≥12 months prior to enrollment. Patients must have a CT or MRI scan of the brain to evaluate for CNS disease within 30 days prior to registration. Patient must not have brain metastases unless: (1) metastases have been treated and have remained controlled for at least two weeks following treatment, AND (2) patient has no residual neurological dysfunction off corticosteroids for at least 1 day. Any radiation therapy completed prior to chemotherapy, except gamma-knife radiosurgery, 1 week prior to chemotherapy.
6. Age >70 years of age at time of signing of the informed consent form.
7. Life expectancy of greater than 12 weeks.
8. ECOG performance status 0-2 (See Appendix A)
9. Patients must have a comprehensive geriatric assessment and chemotherapy toxicity assessment score between 7-17 (See Appendix B, D)
10. Patients must have normal organ and marrow function as defined below:

    * Leukocytes >3,000/mcL
    * ANC > 1,500 cells/mm3Hemoglobin > 9.0g/dL
    * Platelets >100,000 cells/mm3
    * Total bilirubin < 1.5 mg/dL (unless there is a known history of Gilberts Syndrome).
    * AST(SGOT)/ALT(SGPT) ≤2.5 X institutional upper limit of normal
    * Alkaline phosphatase < 2.5 X upper limit of normal in the absence of liver or bone metastasis, or ≤ 5.0 × upper limit of normal range if bone or liver metastases
    * Creatinine clearance >25 mL/min or creatinine <1.5 mg/dL
11. HIV-positive patients on combination antiretroviral therapy are eligible if they have been on ARVs for ≥6 months and undetectable viral loads.
12. Patients must not have documented evidence of acute hepatitis or have an active or uncontrolled infection.
13. No other priormalignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years.
14. Ability to understand and the willingness to sign a written informed consent document in English or a Spanish consent "short form". If language other than English or Spanish, then interpreter will be used to sign English consent form.
15. Patients must have < Grade 2 pre-existing peripheral neuropathy (per CTCAE)

Exclusion Criteria

1. Patients who have had palliative chemotherapy prior to entering the study <12 months from enrollment or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
2. Patients may not be receiving any other investigational agents or have received immunotherapy.
3. Known EGFR or ALK mutated disease (molecular testing not required prior to study entry)
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to carboplatin, or nab-paclitaxel.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Preexisting peripheral neuropathy of Grade 2, 3, or 4 (per Common Terminology Criteria for Adverse Events v4.0)
7. Evidence of active brain metastases, including leptomeningeal involvement (prior evidence of brain metastasis are permitted only if treated and stable and off therapy for ≥ 2 weeks prior to signing Informed consent form. Magnetic Resonance Imaging of the brain (or Computed Tomography scan w/contrast) is preferred for diagnosis.

Min Age: 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rogerio Lilenbaum, MD, Principal Investigator — Yale University
Locations (1):
- Yale Cancer Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Platinum-based Doublet Chemotherapy: * Carboplatin AUC 5 30 minute infusion IV on day 1
  * Nab-paclitaxel 100mg/mg2 30 minute infusion IV on days 1, 8 of a 21 day cycle
  Carboplatin
  Nab-paclitaxel
- Single Agent Chemotherapy: -Nab-paclitaxel 100mg/mg2 30 minute infusion IV on days 1, 8 of a 21 day cycle
  Nab-paclitaxel
Period: Overall Study
Arm/Group | Platinum-based Doublet Chemotherapy | Single Agent Chemotherapy
Started | 1 | 2
Completed | 0 | 0
Not Completed | 1 | 2
Not completed — Death | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Platinum-based Doublet Chemotherapy | Single Agent Chemotherapy | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure-free Survival
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum-based Doublet Chemotherapy | Single Agent Chemotherapy
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

2. Secondary Outcome: Overall Response Rate
Time Frame: start of treatment to disease progression/recurrence, up to 12 months
Population: The study was terminated after only 3 patients were randomized and all 3 did not respond to treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum-based Doublet Chemotherapy | Single Agent Chemotherapy
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

3. Secondary Outcome: Progression-free Survival
Time Frame: start of treatment to disease progression, up to 12 months
Population: The study was terminated after only 3 patients were randomized and all 3 did not respond to treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum-based Doublet Chemotherapy | Single Agent Chemotherapy
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

4. Secondary Outcome: Overall Survival
Time Frame: Up to 12 months
Population: The study was terminated after only 3 patients were randomized and all 3 did not respond to treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum-based Doublet Chemotherapy | Single Agent Chemotherapy
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

5. Secondary Outcome: Grade 3-5 Adverse Events
Description: Adverse events were characterized using Common Terminology Criteria for Adverse Events (CTCAE)
Time Frame: Up to week 13
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum-based Doublet Chemotherapy | Single Agent Chemotherapy
Number analyzed (Participants) | 1 | 2
Participants
  Overall | 0 | 2
  Grade 3 | 0 | 2
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

6. Secondary Outcome: Symptom Assessment (Measured by FACT-L Symptom Assessment Scale)
Description: The FACT-L is measure of symptoms associated with lung cancer. The higher the score, the greater the symptoms. A maximum score of 136 could be obtained.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Platinum-based Doublet Chemotherapy | Single Agent Chemotherapy
Number analyzed (Participants) | 1 | 2
units on a scale | 89 (NA) — Standard deviation is not calculated. | 44 (26.9)

7. Secondary Outcome: Symptom Assessment (Measured by FACT-L Symptom Assessment Scale)
Description: The higher the score, the greater the symptoms. The FACT-L is measure of symptoms associated with lung cancer. The higher the score, the greater the symptoms. A maximum score of 136 could be obtained. Symptoms were measured following 2 21-day cycles of chemotherapy.
Time Frame: week 6
Population: Only 2 patients were assessed at this timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Platinum-based Doublet Chemotherapy | Single Agent Chemotherapy
Number analyzed (Participants) | 0 | 2
units on a scale |  | 60.5 (19.1)

8. Secondary Outcome: Symptom Assessment (Measured by FACT-L Symptom Assessment Scale)
Description: The FACT-L is measure of symptoms associated with lung cancer. The higher the score, the greater the symptoms. Symptoms were measured following 4 21-day cycles of chemotherapy.
Time Frame: week 12
Population: The study was terminated after only 3 patients were randomized and all 3 did not respond to treatment, these data were not collected at week 12
Arm/Group | Platinum-based Doublet Chemotherapy | Single Agent Chemotherapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Single Agent Chemotherapy | Platinum-based Doublet Chemotherapy
All-Cause Mortality (participants affected / at risk) | 2/2 | 1/1
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Agent Chemotherapy (N=2) | Platinum-based Doublet Chemotherapy (N=1)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Edema limbs (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thromboembolic event (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Agent Chemotherapy (N=2) | Platinum-based Doublet Chemotherapy (N=1)
Anemia (Blood and lymphatic system disorders) | 2 (4) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Blood disorder (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Creatinine Increase (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Edema Limbs (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Epistaxis (General disorders) | 1 (1) | 0 (0)
Eye Pain (Eye disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperkalemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 0 (0)
Hypoalbuminemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hypocalcemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hyponatremia (Blood and lymphatic system disorders) | 2 (6) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Insomnia (General disorders) | 2 (3) | 0 (0)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 2 (7) | 0 (0)
Mucositis oral (Infections and infestations) | 1 (1) | 0 (0)
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
White blood cell decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes